CLINICAL TRIAL: NCT00880867
Title: A Phase I Study of Intratumoral Poly-ICLC Plus Low Dose Local Radiation in Low Grade Recurrent B and T Cell Lymphoma
Brief Title: Intratumoral Poly-ICLC Plus Low Dose Local Radiation in Low Grade Recurrent B and T Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Nevada Cancer Institute (Other)
Collaborators: CLL Topics (Unknown)
Responsible Party: Delva Deauna-Limayo, MD, Nevada Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVCI-0838
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: B Cell Lymphoma; T Cell Lymphoma
Keywords: Low Grade Recurrent B and T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, T-Cell | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Poly-ICLC (Experimental): Poly-ICLC plus low dose local radiation.
  Interventions: Drug: Poly-ICLC

INTERVENTIONS:
Drug: Poly-ICLC — An accessible site of disease (lymph node, cutaneous, subcutaneous, etc.) will be selected by the principal investigator. Patients will then receive two doses of low dose irradiation (2 Gy per day) to that single site on days 1 and 2. Intratumorally or peritumorally Poly-ICLC will be dosed on days 3 and 4 by the physician during weeks 1, 2, 3, 4, and 8.
  Other Names: Hiltonol

SUMMARY:
The primary objective of this study is to evaluate the safety of intratumoral Polyinosinicpolycytidylic acid stabilized with polylysine and carboxymethylcellulose (poly-ICLC)(Hiltonol®) in addition to low-dose local radiotherapy for adult patients with low grade lymphomas, including follicular lymphoma, marginal zone lymphoma, small lymphocytic lymphoma, chronic lymphocytic leukemia, and cutaneous T-cell lymphoma. The secondary endpoints are response rate, immune responses, and durability of responses as well as generation of antiinflammatory response at sites of tumor involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age.
2. Patients must have biopsy confirmed low-grade B-cell lymphoma (follicular, marginal zone, or small cell/chronic lymphocytic leukemia) or mycosis fungoides. B-cell lymphoma patients must have failed at least one prior therapy (chemotherapy or immunotherapy) or mycosis fungoides patients failed at least 1 topical or systemic treatment.
3. Patients must have at least one accessible tumor site that can be injected with poly-ICLC.
4. Patients must have measurable disease other than the injection site.
5. Patients must have a Karnofsky performance status of at least 70%.
6. Patients must have adequate hematologic, renal and liver function (i.e., absolute neutrophil count at least 1500/mm3, Platelets at least 100,000/mm3, creatinine no more than 1.7 mg/dl, total bilirubin no more than 1.5 mg/dl, transaminases no more than 4 times above the upper limits of the institutional normal).
7. Patients must be able to provide written informed consent.
8. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test. While animal testing has been negative, the anti-proliferative activity of this experimental drug may theoretically be harmful to the developing fetus or nursing infant.
9. Required washout period for prior therapy:

   * Topical therapy: 2 weeks.
   * Chemotherapy: 4 weeks
   * Radiotherapy: (including phototherapy): 4 weeks 13 of 26
   * Biological therapies: 4 weeks
   * Other investigational therapy: 4 weeks
   * Rituximab: 12 weeks

Exclusion Criteria:

1. Any history of autoimmune or antibody mediated disease including: systemic lupus, erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, autoimmune hemolytic anemia, pure red cell aplasia, but excluding controlled thyroid disease, or the presence of autoantibodies without clinical autoimmune disease.
2. Off nucleoside or bendustine therapy for a minimum of 6 months
3. Prior treatment with Campath
4. Known history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C (active, prior treatment, or both).
5. Patients with active infection or with a fever > 38.5°C within three days prior to the first scheduled treatment.
6. CNS metastases.
7. Prior malignancy (active within 5 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix.
8. Current anticoagulant therapy (ASA no more than 325 mg/day allowed).
9. Significant cardiovascular disease (i.e., NYHA class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
10. Pregnant or lactating.
11. Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Toxicity (DLT) | Days 1 through 4 during weeks 1, 2, 3, 4, and 8

SECONDARY OUTCOMES:
Tumor Response | Weeks 1 through 4, 8, 12, 16, and q3 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Delva Deauna-Limayo, MD, Principal Investigator — Nevada Cancer Institute
Locations (1):
- Nevada Cancer Institute, Las Vegas, Nevada, United States